CLINICAL TRIAL: NCT04438252
Title: Evaluation of Reliability of Impedance Spectroscopy (CarieScan PRO) in Comparison With Digital Radiograph and ICDAS-II in Detection of Occlusal Carious Lesions: Diagnostic Accuracy Study.
Brief Title: Evaluation of Reliability of CarieScan PRO Compared With Digital Radiograph and ICDAS-II in Detection of Carious Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ramadan Abdelkader, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1711
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cariescan pro (Experimental): device for early caries detection
  Interventions: Device: CariScan Pro; Radiation: Digital Radiograpgy
- ICDAS II (Experimental): Index for caries detection
  Interventions: Diagnostic Test: ICDAS II

INTERVENTIONS:
Diagnostic Test: ICDAS II — Index for caries detection
  Arms: ICDAS II
Device: CariScan Pro — Device for early caries detection
  Arms: Cariescan pro
Radiation: Digital Radiograpgy — Device for digital x-ray imaging
  Arms: Cariescan pro

SUMMARY:
The aim of this study is to evaluate the Clinical performance of alternating current impedance spectroscopy (CarieScan PRO) in comparison with digital radiograph and ICDAS-II in detection of occlusal carious lesions.

DETAILED DESCRIPTION:
The visual examination is routinely used for detecting caries in dental clinics and was also used in recent studies comparing the efficacy of various visual aids. It has the benefit that it is quick and easy to perform, does not need expensive equipment, and can be completed without unnecessary radiation or fluorescence (Ismail, et al., 2007). In the current study, ICDAS-II was set as "gold standard" due to validated relationship between its codes and the histological depth of a carious lesion as in many other studies. In addition, several studies have shown good reproducibility and accuracy of ICDAS-II for caries detection in permanent teeth especially caries lesions in the outer half of the enamel (Gugnani, et al., 2010). Bitewing radiographs are used to determine the depth of caries involvement. Most often, bitewing examination is affiliated with the diagnosis of interproximal caries. It is strongly recommended that these radiographs be used in the diagnosis of occlusal caries into dentin (Pitts NB et al., 1991).

ELIGIBILITY:
Inclusion Criteria of teeth:

* Posterior teeth with dark shadow on occlusal surface.
* Vital upper or lower posterior teeth with no signs of irreversible pulpitis.
* Intact contact with opposing teeth.
* Teeth with no previous restorations in other surfaces.

Exclusion criteria of the teeth:

* Periapical pathology or signs of pulpal pathology.
* Tooth hypersensitivity.
* Possible prosthodontic restoration of teeth.
* Heavy occlusion and occlusal contacts or history of bruxism.
* Severe periodontal affection.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 166 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Dental Caries | slow study completion in average of 1 year
  primary occlusal caries

CONTACTS AND LOCATIONS:
Overall Officials: Olfat ElSayed Hassanien, Doctor, Study Director — Cairo University
Locations (1):
- Faculty Of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided